CLINICAL TRIAL: NCT01864278
Title: A Prospective, Global Multicenter, Single Arm Real-World Registry Investigating the Clinical Use and Safety of the LUTONIX Drug Coated PTA Dilatation Catheter
Brief Title: Lutonix Global SFA Registry
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Collaborators: Bard Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CL0004-01
Record Dates: First submitted 2013-05-21; First posted 2013-05-29 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lutonix Drug Coated Balloon: Paclitaxel coated ballooncatheter
  Interventions: Device: Lutonix Drug Coated Balloon

INTERVENTIONS:
Device: Lutonix Drug Coated Balloon — Subject will receive treatment with the Lutonix Drug Coated Balloon

SUMMARY:
The registry will enroll patients with claudication or ischemic rest pain and an angiographically significant lesion in the superficial femoral or popliteal artery. Subjects will be treated with the LUTONIX Drug Coated PTA Dilatation Catheter carrying the CE Mark per current Instructions for Use(IFU) and followed clinically for a minimum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female ≥18 years of age;
* Rutherford Clinical Category ≤ 4;
* Patient is willing to provide 5-year informed consent and comply with the required follow up;
* Stenotic or obstructive vascular lesions of the femoropopliteal artery;
* Lesion(s) can be treated with available LUTONIX Drug Coated PTA Dilatation Catheter device size matrix per current IFU;
* At least one patent native outflow artery to the ankle free from significant lesion (≥50% stenosis) as confirmed by angiography (treatment of outflow disease is NOT permitted; treatment of in-flow disease is permitted prior to treatment with the LUTONIX Drug Coated PTA Dilatation Catheter).

Exclusion Criteria:

* Patient is currently participating in an investigational drug or device study;
* Inability to take recommended medications as stated in the IFU or non-controllable allergy to contrast;
* Pregnant or planning on becoming pregnant or men intending to father a child;
* Rutherford Class > 4
* Known inadequate distal outflow or planned future treatment of vascular disease distal to the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients (global registry)
Sampling Method: Non-Probability Sample
Enrollment: 691 (Actual)
Dates: Start 2012-12; Primary Completion 2015-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Freedom from Target Lesion Revascularization (TLR) | 12 months
  Efficacy: Freedom from TLR at 12 months.
Freedom from Target Vessel Revascularization(TVR), major index limb amputation, and device- and procedure-related death | 30 days
  Safety: Freedom at 30 days from TVR, major index limb amputation, and device- and procedure-related death

CONTACTS AND LOCATIONS:
Locations (23):
- Allgemeines Krankenhaus Wien, Vienna, Austria
- ZNA Campus Middelheim, Antwerp, Belgium
- CHU Le Bocage, Dijon, France
- Germany (5):
  - Karolinen Hospital Huesten, Arnsberg
  - Diakoniewerk Muenchen, München
  - Medinos Kliniken Sonneberg, Sonneberg
  - Kreiskrankenhaus Viechtach, Viechtach
  - Klinikum Weiden, Weiden
- University General Hospital of Patras, Pátrai, Greece
- Italy (4):
  - AO Cardinal Massaia, Asti
  - IRCCS Policlinico San Donato, San Donato Milanese
  - Azienda Ospedaliera della Valtellina e dalla Valchiavenna, Sondalo
  - AO Ordine Mauriziano, Torino
- Poland (3):
  - Szpital Uniwersytecki nr 2 im. Biziel, Bydgoszcz
  - Szpital Kliniczny Przemienienia Panskiego, Poznan
  - Voivodship Specialist Hospital, Torun
- Hospital Clinico Barcelona, Barcelona, Spain
- Kantonsspital Aarau, Aarau, Switzerland
- United Kingdom (5):
  - Royal Liverpool, Liverpool
  - St Thomas' Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Wythenshawe Hospital, Manchester
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Derived] Thieme M, Von Bilderling P, Paetzel C, Karnabatidis D, Perez Delgado J, Lichtenberg M; Lutonix Global SFA Registry Investigators. The 24-Month Results of the Lutonix Global SFA Registry: Worldwide Experience With Lutonix Drug-Coated Balloon. JACC Cardiovasc Interv. 2017 Aug 28;10(16):1682-1690. doi: 10.1016/j.jcin.2017.04.041. Epub 2017 Aug 2. PMID 28780030